CLINICAL TRIAL: NCT05069506
Title: Short-term Effects of Goat Milk Yogurt on Postprandial Glycemic Responses, Arterial Blood Pressure, Energy Intake and Satiety
Brief Title: Effects of Goat Milk Yogurt on Postprandial Glycemic Responses, Arterial Blood Pressure and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor in Nutrition and Metabolism, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HRBD 24 Session 04/04/2019 NHA
Record Dates: First submitted 2019-07-09; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetite; Lack or Loss, Nonorganic Origin
MeSH Terms: interventions — Glucose; Milk; Lactic Acid

STUDY DESIGN:
Intervention Model Description: Other: Glucose as reference food Other: goat milk yogurt as test food Other: goat milk yogurt with currants as test food Other: currants as test food Other: sultanina raisins as test food Other: goat milk preload Other: milk with lactic acid preload
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Glucose as reference food (Experimental): Twelve healthy, normal-weight subjects (male: 4, female: 8) after 10-14 hr fast, consumed 25g available carbohydrate from glucose, three times, in different weeks as reference foods along with 250ml water; and 25g available carbohydrates from a) goat milk yogurt, b) goat milk yogurt and currants, c) currants, d) sultanina raisins, one time each, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Goat milk as test food; Other: Goat milk and currants as test food; Other: Currants as test food; Other: Sultanina raisins as test food; Other: Goat milk yogurt as preload; Other: Milk with lactic acid as preload
- Goat milk as test food (Experimental): Twelve healthy, normal-weight subjects (male: 4, female: 8) after 10-14 hr fast, consumed 25g available carbohydrate from glucose, three times, in different weeks as reference foods along with 250ml water; and 25g available carbohydrates from a) goat milk yogurt, b) goat milk yogurt and currants, c) currants, d) sultanina raisins, one time each, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Goat milk as test food; Other: Goat milk and currants as test food; Other: Currants as test food; Other: Sultanina raisins as test food; Other: Goat milk yogurt as preload; Other: Milk with lactic acid as preload
- Goat milk and currants as test food (Experimental): Twelve healthy, normal-weight subjects (male: 4, female: 8) after 10-14 hr fast, consumed 25g available carbohydrate from glucose, three times, in different weeks as reference foods along with 250ml water; and 25g available carbohydrates from a) goat milk yogurt, b) goat milk yogurt and currants, c) currants, d) sultanina raisins, one time each, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Goat milk as test food; Other: Goat milk and currants as test food; Other: Currants as test food; Other: Sultanina raisins as test food; Other: Goat milk yogurt as preload; Other: Milk with lactic acid as preload
- Currants as test food (Experimental): Twelve healthy, normal-weight subjects (male: 4, female: 8) after 10-14 hr fast, consumed 25g available carbohydrate from glucose, three times, in different weeks as reference foods along with 250ml water; and 25g available carbohydrates from a) goat milk yogurt, b) goat milk yogurt and currants, c) currants, d) sultanina raisins, one time each, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Goat milk as test food; Other: Goat milk and currants as test food; Other: Currants as test food; Other: Sultanina raisins as test food; Other: Goat milk yogurt as preload; Other: Milk with lactic acid as preload
- Sultanina raisins as test food (Experimental): Twelve healthy, normal-weight subjects (male: 4, female: 8) after 10-14 hr fast, consumed 25g available carbohydrate from glucose, three times, in different weeks as reference foods along with 250ml water; and 25g available carbohydrates from a) goat milk yogurt, b) goat milk yogurt and currants, c) currants, d) sultanina raisins, one time each, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Goat milk as test food; Other: Goat milk and currants as test food; Other: Currants as test food; Other: Sultanina raisins as test food; Other: Goat milk yogurt as preload; Other: Milk with lactic acid as preload
- Goat milk as preload (Experimental): Forty-five healthy subjects (male: 12, female: 33) were offered a standardized breakfast and 2h after consumed one of the two preloads (goat milk yogurt and milk with lactic acid) served as snack in random order. Three hours after, subjects were given ad libitum access to a meal (lunch and dessert). Foods were weighed at the time of serving and any leftovers were weighed again after meal to determine the amount of food consumed. Fingertip capillary blood glucose samples were collected before and after foods. Subjective appetite ratings were collected using 100mm visual analogue scales (VAS).
  Interventions: Other: Glucose as reference food; Other: Goat milk as test food; Other: Goat milk and currants as test food; Other: Currants as test food; Other: Sultanina raisins as test food; Other: Goat milk yogurt as preload; Other: Milk with lactic acid as preload
- Milk with lactic acid as preload (Experimental): Forty-five healthy subjects (male: 12, female: 33) were offered a standardized breakfast and 2h after consumed one of the two preloads (goat milk yogurt and milk with lactic acid) served as snack in random order. Three hours after, subjects were given ad libitum access to a meal (lunch and dessert). Foods were weighed at the time of serving and any leftovers were weighed again after meal to determine the amount of food consumed. Fingertip capillary blood glucose samples were collected before and after foods. Subjective appetite ratings were collected using 100mm visual analogue scales (VAS).
  Interventions: Other: Glucose as reference food; Other: Goat milk as test food; Other: Goat milk and currants as test food; Other: Currants as test food; Other: Sultanina raisins as test food; Other: Goat milk yogurt as preload; Other: Milk with lactic acid as preload

INTERVENTIONS:
Other: Glucose as reference food — Twelve subjects (male: 4 female: 8) consumed 25g glucose diluted in 150ml water, two times, in different weeks, within 5-10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
Other: Goat milk as test food — Twelve subjects (male: 4 female: 8) consumed 617 g goat milk yogurt, offering 25g available carbohydrate along with 250 mL water, one time, in different weeks, within 10-15 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
Other: Goat milk and currants as test food — Twelve subjects (male: 4 female: 8) consumed 308 g goat milk yogurt and 19 g currants, offering 25g available carbohydrate along with 250 mL water, one time, in different weeks, within 10-15 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
Other: Currants as test food — Twelve subjects (male: 4 female: 8) consumed 37.8 g currants, offering 25g available carbohydrate along with 250 mL water, one time, in different weeks, within 10-15 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
Other: Sultanina raisins as test food — Twelve subjects (male: 4 female: 8) consumed 37.5 g sultanina raisins, offering 25g available carbohydrate along with 250 mL water, one time, in different weeks, within 10-15 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
Other: Goat milk yogurt as preload — Forty-five healthy subjects (male: 12, female: 33) consumed a standardized breakfast (bread and honey) and 2h after were offered a preload given as snack (200g goat milk yogurt). Three hours after, subjects were given ad libitum access to a meal (lunch and dessert). The meal consisted of rice, roasted chicken breast and chocolate vanilla cake. Foods were weighed before serving and any leftovers were weighed again after meal. Fingertip capillary blood glucose samples were taken before breakfast, 120min after breakfast; before preload, 120minand 180minpost-preload consumption; before meal (lunch and dessert), 60minand 120min post-meal consumption. Subjective appetite ratings were assessed with 100mm VAS.
Other: Milk with lactic acid as preload — Forty-five healthy subjects (male: 12, female: 33) consumed a standardized breakfast (bread and honey) and 2h after were offered a preload given as snack (200g milk with lactic acid). Three hours after, subjects were given ad libitum access to a meal (lunch and dessert). The meal consisted of rice, roasted chicken breast and chocolate vanilla cake. Foods were weighed before serving and any leftovers were weighed again after meal. Fingertip capillary blood glucose samples were taken before breakfast, 120min after breakfast; before preload, 120minand 180minpost-preload consumption; before meal (lunch and dessert), 60minand 120min post-meal consumption. Subjective appetite ratings were assessed with 100mm VAS.

SUMMARY:
This study investigated any potential associations between two preloads offered as snacks and postprandial glycemic response, subjective appetite and energy intake in healthy, normal weight adults

DETAILED DESCRIPTION:
This study aimed at 1. firstly determine the glycemic index (GI) of a) goat milk yogurt b) goat milk yogurt with currants, c) currants and d) sultanina raisins, all containing 25 gr available carbohydrates and 2. test the hypothesis that a goat milk yogurt consumed as a snack before a meal, compared to milk with lactic acid would: a) have greater short-term effect on satiety measured by subsequent ad libitum meal intake, b) induce greater satiety as assessed by visual analogue scales (VAS) and c) reduce postprandial glycemic response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, non-diabetic men and women individuals with normal body mass index (BMI; between 18.5 and 24.9 kg/m2)

Exclusion Criteria:

* Severe chronic disease (e.g. tumors, manifest coronary heart disease, diabetes mellitus, severe kidney or liver conditions, endocrine and immunological conditions)
* Gastrointestinal disorders (e.g. chronic inflammatory bowel disease)
* Lactose intolerance
* Pregnancy
* Competitive sports
* Lactation
* Alcohol
* Drug dependency

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose | 7 hours
  Clinically useful change in serum glucose (mg/dL), defined as the restoration of glucose within normal limits during the 2hr glucose tolerance test and for a total of 5 hours

SECONDARY OUTCOMES:
Subjective appetite ratings | 7 hours
  Useful change in subjective appetite (hunger, desire to eat, motivation to eat, preoccupation with thoughts of food, thirst) scores 0 up to 10 from 100mm Visual Analogue Scales
Energy intake after preload | 6 hours
  Useful change in energy intake (kcal) the day of the intervention (actual weighing of foods in grams consumed and leftovers using a Kern & Sohn (Germany) food weight scale (Max 3500 g, d=0.01g) and analysis from 24hr recalls using Diet Analysis Software
Arterial blood pressure | 7 hours
  Clinically useful change in systolic and diastolic blood pressure (mmHg) before and after consumption of test foods

CONTACTS AND LOCATIONS:
Locations (1):
- Agricultural University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No